CLINICAL TRIAL: NCT05054439
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of SI-B001 in Combination With Paclitaxel in the Treatment of Recurrent and Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Clinical Study of SI-B001 in Combination With Paclitaxel in the Treatment of Recurrent and Metastatic HNSCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001_206
Record Dates: First submitted 2021-08-22; First posted 2021-09-23 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SI-B001 combined with paclitaxel (Experimental): SI-B001 in combination with paclitaxel for the treatment of recurrent metastatic head and neck squamous cell carcinoma (non-nasopharyngeal carcinoma) with disease progression or intolerance.； The patient had previously received anti-PD-1 mab ± platinum-based chemotherapy； Patients' previous treatment line should be ≤2L.
  Interventions: Drug: SI-B001; Drug: Paclitaxel

INTERVENTIONS:
Drug: SI-B001 — Si-b001 is administered by intravenous drip once a week (QW). The first intravenous infusion is 120 min±10min. If the infusion reaction can be tolerated during the first infusion, the subsequent infusion can be completed in 60-120 min.
Drug: Paclitaxel — The dosage of paclitaxel was 80mg/m2 QW. SI-B001 and paclitaxel were used on the same day. After SI-B001 infusion, paclitaxel was pretreated and injected for no less than 3 hours.

SUMMARY:
This multi-center, open label phase II clinical study is performed in patients with relapsed metastatic head and neck squamous cell carcinoma (non-nasopharyngeal carcinoma) progressed on prior 1st or 2nd line with anti-PD-1 mab ± platinum-based chemotherapy. This study is investigating the safety and efficacy of SI-B001 at optimal combination dose with paclitaxel in patients.

ELIGIBILITY:
Inclusion Criteria:

1. The participants could understand and sign the informed consent form and must participate voluntarily.
2. No gender limit;
3. Age: ≥18 years old
4. Locally advanced squamous cell carcinoma of the head and neck confirmed by histology or pathology as recurrent metastatic or without indications of radical local treatment;
5. Patients who failed or were intolerant to previous anti-PD-1 monoclonal antibody, platinum-containing chemotherapy or anti-PD-1 monoclonal antibody monotherapy Treatment failure of PD-1 refers to disease progression during or after PD-1 treatment;

   Failure of platinum-containing chemotherapy refers to:
   1. disease progression during or after platinum-containing chemotherapy;
   2. recurrence or disease progression within 6 months of platinum-containing multi-mode therapy;
6. Previously received only ≤ 2-line treatment for recurrent and metastatic squamous cell carcinoma of the head and neck;
7. Agree to provide tumor tissue samples (FFPE block or 10 unstained sections of 5μm size) or fresh tissue samples that have been archival within 1 year of primary or metastatic lesion. If the patient fails to provide them, they can be included after the investigator's judgment;
8. There must be at least one measurable lesion in accordance with the RECIST V1.1 definition. Tumor lesions located in the area of previous radiotherapy or other local regional treatment sites are generally not measurable unless there is definite progression of the lesion or the lesion persists three months after radiotherapy;
9. Physical fitness ECOG score 0 or 1;
10. Toxicity of previous antitumor therapy has returned to ≤1 as defined by NCI-CTCAE V5.0 (except for toxicity that the investigators judged to be of no safety risk, such as hair loss, grade 2 peripheral neurotoxicity, and stabilized hypothyroidism after hormone replacement therapy);
11. Organ function levels must meet the following requirements and meet the following standards:

    1. Bone marrow function: absolute neutrophil count (ANC)≥1.5×10*9/L, platelet count ≥100×10*9/L, hemoglobin ≥90 g/L;
    2. Liver function: Total bilirubin TBIL≤1.5×ULN (total bilirubin ≤3×ULN in Subjects with Gilbert's syndrome, liver cancer or liver metastasis), AST and ALT ≤2.5×ULN in patients without liver metastasis, AST and ALT ≤5.0×ULN in patients with liver metastasis;
    3. Renal function: creatinine (Cr) ≤1.5×ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula);
    4. Urine routine / 24-hour protein quantification: qualitative urine protein ≤1+ (if qualitative urine protein ≥2+, 24-hour protein < 1g can be included in the group);
    5. Cardiac function: left ventricular ejection fraction ≥50%;
    6. Coagulation function: International standardized ratio (INR) ≤1.5×ULN, and activated partial thrombin time (APTT) ≤1.5×ULN;
12. Eligible patients (male and female) who are fertile must agree to use a reliable contraceptive method (hormonal or barrier method or abstinence, etc.) with their partner during the trial and for at least 6 months after the last medication; women of childbearing age must have a negative blood or urine pregnancy test within 7 days prior to the first use of the study drug.

Exclusion Criteria:

1. Squamous cell carcinoma with primary site of nasopharynx or skin;
2. Have received chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor therapy within 4 weeks prior to the first use of the study drug, except the following:

   * Nitrosorea or mitomycin C within 6 weeks before the first administration of the study drug;
   * Oral fluorouracil and small molecule targeted drugs are 2 weeks before the first administration of the study drug or within the 5 half-lives of the drug (whichever is longer);
   * The traditional Chinese medicines with anti-tumor indications were within 2 weeks before the first use of the study drug;
3. Received an unmarketed clinical investigational drug or treatment within 4 weeks prior to the first use of the investigational drug;
4. Has undergone major organ surgery (excluding needle biopsy, tracheotomy, gastrostomy, etc.) or has significant trauma within 4 weeks before the first use of study drugs, or needs to undergo elective surgery during the trial;
5. Patients with prior use of paclitaxel or albumin paclitaxel or paclitaxel liposome;
6. Previous recipients of allogeneic hematopoietic stem cell transplantation or organ transplantation;
7. A history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

   * Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, grade iii atrioventricular block, etc.
   * In the resting state, QT interval was prolonged (QTc > 450 msec in men or QTc > 470 msec in women).
   * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grades 3 or higher cardio-cerebrovascular events within 6 months prior to the first administration;
   * New York Heart Association (NYHA) heart function grade ≥II heart failure;
8. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, systemic treatment of psoriasis, rheumatoid arthritis, inflammatory bowel disease, and Hashimoto's thyroiditis, etc., with the exception of type I diabetes, only replacement therapy can control hypothyroidism, no systemic treatment of skin disease (e.g., vitiligo, psoriasis);
9. A history of other malignancies within 5 years prior to first administration, except for radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or radical excised carcinoma in place, and second primary squamous cell carcinoma of the head and neck;
10. Poorly controlled hypertension (systolic blood pressure & GT; 150 mmHg or diastolic pressure > 100 mmHg);
11. Pulmonary disease defined as grade 3 or higher according to CTCAE V5.0; Patients with past or present interstitial lung disease (ILD);
12. Cerebral parenchymal or meningeal metastases with clinical symptoms are not suitable for inclusion by the investigator;
13. Experienced ≥ grade 3 infusion-related reactions during previous anti-EGFR antibody therapy;
14. Known allergies to paclitaxel or its standard pretreatments or other contraindications to products containing castor oil;
15. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > 104) or hepatitis C virus infection (HCV-RNA > center detection lower limit);
16. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.;
17. Pregnant or lactating women;
18. Persons with mental disorders or poor compliance;
19. The investigator considers that the subject has a history of other serious systemic diseases or other reasons and is not suitable to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 2 years
  (Objective Response Rate )

SECONDARY OUTCOMES:
Tmax | Up to 2 weeks
  Time to maximum serum concentration
PFS | Up to 2 years
  Progression-free Survival
DCR | Up to 2 years
  Disease Control Rate
OS | Up to 2 years
  overall survival
TEAE | Up to 2 years
  Treatment Emergent Adverse Events
Cmax | Up to 2 years
  maximum serum concentration
Ctrough | Up to 2 years
  Minimum serum concentration
ADA | Up to 2 years
  anti-SI-B001 antibody

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Union Hospital Tongji Medical College， Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang